CLINICAL TRIAL: NCT00286403
Title: Combination Fenoldopam Mesylate and Intravenous MESNA (2-mercaptoethane Sulphonate)in Early Acute Kidney Injury (AKD): A Randomized, Double-Blind Placebo Controlled Clinical Trial
Brief Title: Vasodilators and Anti-Oxidant Therapy in Early ATN
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to logistics at a local hospital.
Sponsor: Southeast Renal Research Institute (Other)
Collaborators: Dialysis Clinic, Inc. (Industry)
Responsible Party: James A. Tumlin, MD, Southeast Renal Research Institute
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MCAT-1
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Acute Renal Failure
Keywords: Acute Tubular Necrosis; antioxidants; Fenoldopam
MeSH Terms: conditions — Acute Kidney Injury; Kidney Cortex Necrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fenoldopam Mesylate and/or MESNA

SUMMARY:
Patients developing kidney failure after open heart surgery experience an abrupt decrease in blood flow to the kidney. The investigators hypothesize that administration of fenoldopam mesylate (a drug that increases blood flow to the kidney) to patients early in the course of their disease could reduce progression to dialysis-dependent acute renal failure. The investigators also hypothesize that restoring blood flow could induce additional injury to the kidney through the release of reactive oxygen species. Therefore, patients in this protocol will be randomized to receive a fenoldopam or the anti-oxidant MESNA. The investigators hypothesize that combination treatment with Fenoldopam and MESNA will decrease the incidence of death or dialysis at 21 days in patients with early post-operative acute renal failure.

DETAILED DESCRIPTION:
Primary Hypotheses:

* Combination therapy with intravenous fenoldopam mesylate and MESNA will reduce the incidence of dialysis and all cause mortality at 21 days in patients with established acute tubular necrosis (ATN).
* The combination of fenoldopam mesylate and Intravenous MESNA reduces the level of reactive oxygen species released following restoration of renal blood flow in patients with ischemic ATN.

Specific Aims

1. To conduct a multicenter, double blind, trial comparing the efficacy of a 72-hour infusion of fenoldopam mesylate or combination of fenoldopam plus intravenous MESNA to reduce the incidence of dialysis or all-cause mortality at 21 days in patients with ischemic ATN.
2. To determine the effects of fenoldopam mesylate alone or in combination with MESNA on reperfusion injury as evidenced by changes in the level of urinary 15-F2t-isoprostanes The rational is that failure of parenteral vasodilators to reduce the incidence of death or dialysis among patients with ATN may involve the extension of tubular injury through normalization of renal blood flow and subsequent reperfusion injury. Moreover, the generation of reactive oxidative species in areas of hypoxia could blunt impair regional blood flow in the kidney through inhibition of nitric oxide production.
3. To serially measure the urinary content of ICAM-1, VCAM-1, KIM-1, P-selectin, E-selectin, MCP-1and Cyr-61 and determine the ability of specific markers to identify patients progressing to dialysis dependent ATN.

The rational is that ICAM-1 is expressed by ischemic endothelium and facilitates neutrophile migration into areas of necrotic epithelium. We will determine whether rising urinary ICAM-1 will identify patients with progressive dialysis-dependent ATN. Specific aim #3 will also examine whether a reduction in dialysis or all cause mortality by fenoldopam mesylate correlates with reduced urinary expression of ICAM-1 or other cell adhesion molecules. The serum, plasma, urine supernatant and urinary casts obtained from patients enrolled in this trial will be made available to other investigators involved in the study of early ATN.

ELIGIBILITY:
Inclusion Criteria:

* Post-operative patients with serum creatinine (Cr) rising 0.3 mg/dl or more than 25% above admission levels within a single 24-hour period will be considered eligible.
* Central Venous Access: [CVP > 6 cm H2O without mechanical ventilation] [CVP > 9 cm H2O with mechanical ventilation]
* Mean arterial pressure > 70 mm Hg receiving up to two vasopressors including:

  * Nor-epinephrine (0.01-1.5g/kg/min)
  * Phenylephrine (0.1-7.0g/kg/min
  * Vasopressin (0.1-1.5 mU/kg/min)

Exclusion Criteria:

* Patients with APACHE scores greater than 30 (or felt by the principal investigators to be unlikely survive more than 24 hours).
* Patients requiring 3 or more presser agents to maintain a MAP of 70 mm Hg or greater.
* Patients on two vasopressors with a MAP < 70 mm Hg will not be considered for enrollment
* Patient with baseline serum Cr > 3.0 mg/dl
* Patients with known bacteremia and/or the Systemic Inflammatory Response Syndrome (SIRS)
* Patients ATN secondary to aminoglycosides or amphotericin B or equivalent anti-fungal drug
* Patients on chronic peritoneal or hemodialysis
* Patients receiving acute peritoneal or hemodialysis during current hospitalization
* Patients on dopamine infusion within the previous 12 hours
* Patients with known HIV seropositivity and past history of opportunistic infection
* Pregnant or lactating women
* Patients with history of uncontrolled atrial or ventricular cardiac arrhythmia
* Patients under the influence of alcohol or other drugs
* Patients enrolled in a previous investigational study within15 days of enrollment
* Patients with a known hypersensitivity to fenoldopam mesylate
* Patients with a known history of glaucoma.
* Patients with cirrhosis of the liver and/or portal hypertension
* Patients with toxic levels of calcineurin inhibitors (FK-506 or CsA) or acute allograft rejection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Death or Dialysis at 21 days

SECONDARY OUTCOMES:
Peak serum Cr and Duration of ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: James A Tumlin, MD, Principal Investigator — Southeast Renal Research Institute; Micheal Kutner, Ph.D., Study Director — Rollins School Public Health
Locations (2):
- United States (2):
  - Chawala, M. MD, Washington D.C., District of Columbia
  - Mandeep Grewal, Chattanooga, Tennessee

REFERENCES:
- [Background] Tumlin JA, Finkel KW, Murray PT, Samuels J, Cotsonis G, Shaw AD. Fenoldopam mesylate in early acute tubular necrosis: a randomized, double-blind, placebo-controlled clinical trial. Am J Kidney Dis. 2005 Jul;46(1):26-34. doi: 10.1053/j.ajkd.2005.04.002. PMID 15983954
- [Derived] Esezobor CI, Bhatt GC, Effa EE, Hodson EM. Fenoldopam for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD012905. doi: 10.1002/14651858.CD012905.pub2. PMID 39607014